CLINICAL TRIAL: NCT03328208
Title: Nonpharmacologic Reduction of Periprocedural Pain, Anxiety, and Prescription Drug Use
Brief Title: Nonpharmacologic Reduction of Periprocedural Distress and Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hypnalgesics, LLC (Industry)
Collaborators: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R43AT009517 (NIH)
Record Dates: First submitted 2017-10-21; First posted 2017-11-01 (Actual); Results first posted 2020-03-04 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Dental Anxiety; Dental Pain; Drug Use; Opioid Use
Keywords: Nonpharmacologic analgesia; Medical app; Relaxation
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Intervention Model Description: This is a single-blind placebo-controlled trial comparing a Comfort Talk® calmative app (App Group) with a white noise app (Control Group).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The four tablets used in the study will be labeled A,B,C,D and will be preloaded with the app or white noise by the Hypnalgesics, LLC in randomized sequence. Personnel at TUSDM will not be aware which tablet presents test or control content. The opening screen and option screen of the white noise control app will use the same color scheme and lay-out as the one of the test Comfort Talk app. The statistical team will receive the encoded data entries and will not be informed about the content of the tablets until all analyses are completed. Since they also will not have direct contact with the study patients they are also not at risk of becoming unblinded during app use by the patients.
  At the end of their visit, patients will receive a sealed envelope which according to their number will either contain a download coupon for the app for home use or a thank you note. To maintain blinding, all patients who send their diaries back will receive a download coupon.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comfort Talk® App Group (Experimental): Patients will receive a tablet preloaded with the Comfort Talk® app in the dental waiting room on an intent-to-treat basis. They can listen as much or as little as they wish during waiting and during their dental treatment. Upon departure, they will receive a download coupon for the app for home use.
  Interventions: Other: Comfort Talk® app
- White Noise Group (Active Comparator): Patients will receive a tablet preloaded with a white noise app in the dental waiting room on an intent-to-treat basis. They can listen as much or as little as they wish during waiting and during their dental treatment.
  Interventions: Other: White Noise app

INTERVENTIONS:
Other: Comfort Talk® app — Test app
  Other Names: Relaxation app
  Arms: Comfort Talk® App Group
Other: White Noise app — White Noise app built to mimic appearance of Comfort Talk® test app
  Other Names: Control app
  Arms: White Noise Group

SUMMARY:
Objectives of this Phase I pilot trial are to provide data towards assessing and facilitating feasibility of a larger scale Phase II trial in which the effects of a calmative Comfort Talk® app can be unequivocally evaluated.

Towards this goal we will pursue following outcome parameters for

Phase I: Feasibility/acceptability assessment:

Primary outcome parameter:

• ability to obtain complete on-site data sets from at least 90% of patients enrolled (with at least 40% from patients in the app group and at least 40% from patients in the control group).

Secondary outcome parameters:

* ability to enroll 60 patients by day 150 after initiation of recruitment in the clinic (=day 1)
* obtain 38 packages of filled out diary cards (at least 16 from patients in the app group and at least 16 from patients in the control group)
* 90% of patients in app group listen to app ≥5 min

Phase II preparation primary outcome parameter

• anxiety at the end of the waiting room time

Secondary outcome parameters

* pain the end of the waiting room time
* anxiety during treatment
* pain during treatment
* anxiety during 1 week after treatment
* pain during 1 week after treatment
* use of units of sedatives and analgesics during 1 week after treatment (assessed by prescription at end of the visit)
* patient satisfaction

DETAILED DESCRIPTION:
The design is a single-blind, placebo controlled clinical trial to test the feasibility of the trial design assessing the ability of a Comfort Talk® app to nonpharmacologically reduce anxiety, pain, and periprocedural drug use in individuals 18 years of age and older undergoing outpatient treatment in the Craniofacial Pain Center of the Tufts School of Dental Medicine.

The trial is a single-site pilot trial to assist in sample size estimation in a pivotal trial to test the hypothesis that listening to a Comfort Talk® app with calmative content reduces pain, anxiety, and post-procedural medication use.

Eligible patients at the Craniofacial Pain Center at the Tufts School of Dental Medicine (TUSDM) will be randomized to listen to a tablet containing a calmative Comfort Talk® app or app with white noise on an intent-to-treat basis. Their anxiety and pain measures will be recorded on validated 0-10 scales and before listening, at the end of the waiting room period, and every 10 minutes while on the dental chair.

All patients will be given a packet with diary cards to record their levels of anxiety, pain, and drug use daily for 7 days after their visit and asked to send those back. Subjects will be mailed a $25 check upon returning their diaries.

Patients randomized to the Comfort Talk® app will receive a download coupon for the app before leaving TUSDM, those randomized to the control condition (white noise) will receive a download coupon after they send in their diary cards.

Interventions and Duration

Approximately 1 hour and 15 minutes (Up to 30 minutes more than the scheduled standard of care visit, which will typically last up to 45 minutes):

Patient will be asked to come in ½ hour early before an already scheduled appointment. They will be taken to a private area, report their demographics, and if eligible consented and fill out a NIDA Quick Screen.

The participant will then be verbally asked to indicate his/her pain and anxiety levels on validated 0-10 scales. The research assistant will then hand the participant a tablet containing, depending on the group attribution, either the app (App Group) or white noise (Control Group) and will be shown how to operate the tablet.

Participant will then return to the clinic waiting area with the tablet and wait for their regularly scheduled appointment. The patient will be at liberty to when and for how long to listen. At the end of the waiting room period the participant will be queried again for their levels of pain and anxiety.

After the participant enters the treatment room, he or she will be able to continue to listen to the app or white noise on the tablet. The research assistant will ask the participant every 10 min to indicate their pain and anxiety levels. The research assistant will note the duration of chair time, the amount of lidocaine given, if any or which other medications were given during the appointment, and whether the dental practitioner prescribed opioid, prescription or non-prescription drugs at the end of the visit.

Before leaving home, the participant will be asked to fill out a satisfaction survey based on a modified Press Ganey Template. The participant will then receive a diary card on which to note pain, average and maximal pain as well its location, use of non-prescription, prescription, and opiate drugs, use of the app, and be provided pre-stamped envelopes. Patients will be asked to complete the diary daily before bedtime for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a dental procedure at the Craniofacial Pain Center
* Able to hear, write and read in English, as the ComfortTalk® scripts, study scales and take-home diary are in English
* Able to operate a standard smart tablet or smart phone and have access to a smart tablet, smart phone at home, or computer-based app download
* Willing and able to give informed consent

Exclusion Criteria:

* Known acute psychiatric disorder, such as multiple personalities which will be assessed on the medical history form
* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira V Lang, MD, PhD, Principal Investigator — Hypnalgesics, LLC
Locations (2):
- United States (2):
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - Hypnalgesics, LLC, Brookline, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Comfort Talk® App Group | White Noise Group
Started | 37 | 35
Completed | 37 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comfort Talk® App Group | White Noise Group | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 27 | 58
  >=65 years | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 21 | 50
  Male | 8 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 34 | 71
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 31 | 30 | 61
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 37 | 35 | 72
Pain [Mean (Full Range); unit: units on a scale] — Self-reported pain on a verbal scale with 0=no pain at all and 10=worst pain possible at the beginning of the waiting room time
  units on a scale | 3.4 [0 to 9] | 2.8 [0 to 9] | 3.1 [0 to 9]
Anxiety [Mean (Full Range); unit: units on a scale] — Self-reported anxiety on a verbal scale with 0=no anxiety at all and 10=worst anxiety possible at the beginning of the waiting room time
  units on a scale | 2.6 [0 to 7] | 2.5 [0 to 9] | 2.6 [0 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete On-Site Data Sets
Description: Feasibility defined as the ability to obtain complete on-site data sets from at least 90% of participants enrolled (with at least 40% from patients in the app group and at least 40% from patients in the control group).
Time Frame: Duration of outpatient clinic visit (up to 2 hrs)
Population: Participants enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 37 | 35
Participants | 37 | 35

2. Secondary Outcome: Number of Days to Enroll 60 Participants
Description: Feasibility measure defined as the ability to enroll 60 participants by day 150 after initiation of recruitment in the clinic (=day 1). Outcome measure are numbers of office days from the start of enrollment
Time Frame: Up to 150 days
Population: Number of participants within the cohort of the first 60 participants
Measure: Number; unit: Days
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 31 | 29
Days | 106 | 106

3. Secondary Outcome: Number of Participants Returning Diary Card Packages
Description: Follow-up feasibility defined as obtaining 38 packages of filled out diary cards (at least 16 from patients in the app group and at least 16 from patients in the control group)
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 37 | 35
Participants | 15 | 11

4. Other Pre Specified Outcome: Anxiety at the End of the Waiting Room Time (Change as Compared to Beginning of the Waiting Room Time)
Description: Anxiety as measured by self-report on a 0-10 scale with 0=no anxiety at all and 10=worst anxiety possible; change from the beginning to the end of the waiting room time
Time Frame: Up to 60 min
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 37 | 35
units on a scale | -0.81 [-1.21 to -0.41] | -0.66 [-1.16 to 0.16]
Statistical Analysis 1: Comparison: Comfort Talk® App Group vs White Noise Group; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.724

5. Other Pre Specified Outcome: Pain the End of the Waiting Room Time (Change as Compared to Beginning of the Waiting Room Time)
Description: Pain as measured by self-report on a 0-10 scale with 0=no pain at all and 10=worst pain possible; change from the beginning to the end of the waiting room time
Time Frame: Up to 60 min
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 37 | 35
units on a scale | -0.76 [-1.15 to -0.37] | -0.26 [-0.56 to -0.05]
Statistical Analysis 1: Comparison: Comfort Talk® App Group vs White Noise Group; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.038

6. Other Pre Specified Outcome: Pain During Dental Treatment
Description: Time course of pain as measured by self-report on a 0-10 scale with 0=no pain at all and 10=worst pain possible (average over 10 minute intervals)
Time Frame: Up to 120 min
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 37 | 35
units on a scale | 2.5 (2.0) | 2.5 (1.9)

7. Other Pre Specified Outcome: Anxiety During Dental Treatment
Description: Time course of anxiety as measured by self-report on a 0-10 scale with 0=no anxiety at all and 10=worst anxiety possible (average over 10 minute intervals)
Time Frame: Up to 120 min
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 37 | 35
units on a scale | 2.2 (2.1) | 2.0 (1.7)

8. Other Pre Specified Outcome: Average Maximal Anxiety During 1 Week After Dental Treatment
Description: Average maximal daily anxiety as measured daily by self-report on a 0-10 scale with 0=no anxiety at all and 10=worst anxiety possible
Time Frame: 7 days
Population: Participants who returned their diary card packages
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 15 | 11
units on a scale | 2.3 (1.7) | 2.3 (1.9)

9. Other Pre Specified Outcome: Average Maximal Pain During 1 Week After Treatment
Description: Average of maximal daily pain as measured daily by self-report on a 0-10 scale with 0=no pain at all and 10=worst pain possible
Time Frame: 7 days
Population: Participants who returned their diary card packages
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 15 | 11
units on a scale | 2.9 (1.4) | 3.1 (1.2)

10. Other Pre Specified Outcome: Number of Participants Receiving New Prescriptions for Drugs
Description: Participants receiving new prescriptions for drugs at the end of their visit for the subsequent week (alone or in combination opioids, non-opioid analgesics, anxiolytics, muscle relaxants, triptan, and/or anticonvulsants)
Time Frame: 7 days
Population: All enrolled participants
Measure: Number; unit: participants
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 37 | 35
participants | 8 | 5

11. Other Pre Specified Outcome: Patient Satisfaction
Description: Patient satisfaction on a questionnaire at the end of the outpatient clinic visit, modeled after Press Ganey and averaged over 7 domains and groups. Assessment on Likert Scales from 1 (worst)-5 (best)
Time Frame: Up to 3 hrs
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Comfort Talk® App Group | White Noise Group
Number analyzed (Participants) | 37 | 35
units on a scale | 4.6 [3.5 to 5.0] | 4.6 [3.3 to 5.0]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Comfort Talk® App Group | White Noise Group
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 0/37 | 0/35

LIMITATIONS AND CAVEATS:
This was a feasibility study and as such was not powered to find differences in all domains.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03328208/Prot_SAP_000.pdf